CLINICAL TRIAL: NCT03223441
Title: Pulse Wave Velocity as a Predictor for Postoperative Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: Kenichi Ueda (Other)
Responsible Party: Sponsor-Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201502761
Record Dates: First submitted 2017-07-01; First posted 2017-07-21 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Post-Op Complication; Arterial Stiffness
Keywords: Pulse wave velocity; anesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vascular stiffness increases as a person ages, due to the repetitive stress that is put on the vascular system which causes changes in the elasticity of the vessel walls. The increased stiffness of the arteries puts added stress on the circulatory system. This rise in stiffness has been shown to be associated with an increased risk of cardiovascular events, in both presumably healthy patients, as well as elderly patients The current method for assessing perioperative cardiac risk is the Goldman's Revised Cardiac Risk Index (RCRI). This method, however, does not include a direct measurement of arterial stiffness. Applanation tonometry is a non-invasive technique that has been shown to reliably provide indices of arterial stiffness While the use of applanation tonometry has been widely studied in general medicine, it is has not been studied for pre-operative risk assessment in surgical patients.

The purpose of this investigation is to examine whether aortic stiffness is an independent risk factor for developing cardiovascular related adverse events in patients who are having major surgery under general anesthesia.

Applanation tonometry will be performed on the right carotid and femoral arteries to assess carotid-femoral pulse wave velocity, a surrogate for aortic stiffness. (SphygmoCor system, AtCor Medical, Sydney, Australia). The measurement will be obtained before induction of general anesthesia in the presurgical area. Patients' medical history, intraoperative hemodynamics, and any postoperative complications will be recorded to determine significant correlations and relationships. This information will potentially help identify future patients that might be at greater risk of developing an adverse cardiovascular event following their surgical procedure.

DETAILED DESCRIPTION:
Background: In 1894 William Osler, MD, said: "You are as old as your arteries." A number of recent studies have confirmed this prescient proclamation. Vascular rather than chronological age is the best predictor of adverse cardiovascular events and mortality from coronary insufficiency, ischemia, myocardial infarction, heart failure, cerebrovascular insufficiency or stroke, and renal insufficiency or failure. We believe it is likely this also applies to perioperative risk of cardiovascular complications from the numerous stress factors associated with major surgery.

Vascular aging leads to central aortic dilation, arterial wall thickening of the media and adventitia with sclerotic changes and increased vascular stiffness. These changes lead to central blood pressure (BP) augmentation, elevated systolic and pulse pressure, along with lowered diastolic BP. (1) Central more elastic vessels cushion and dampen pressure oscillations with left ventricular (LV) ejection and transfer this stored energy into continuing antegrade pulse waves along the arterial tree during diastole. (2) the pulse wave is also reflected back centrally when it meets higher flow resistance at major artery branch points and muscular arteries resulting in central aortic combination wave. In a younger compliant central aorta the reflected waves arrive after aortic valve closure, augmenting early diastolic perfusion pressure an coronary blood flow. Elderly stiff aorta and major arteries vessels transfer both antegrade and retrograde pulse waves faster. If heart rate is slow enough an asystole long enough, this combination wave will arrive at the central aorta during late systole. This elevates LV workload, resulting in compensatory left ventricular hypertrophy (LVH). In addition, disappearance of the diastolic combination wave lowers coronary perfusion pressure, increasing the risk of coronary insufficiency for the hypertrophied LV wall.

Unfortunately, high blood flow coronary, and renal arteries are not so muscular that they can reduce the impact of high combination systolic pressure waveforms. This induces chronic kinetic injury to these high blood flow vessels and organs. Increased pulsatility leads to arterial remodeling and microcirculation damage in brain and kidney, small lacunare infarcts, white matter lesions associated with cognitive dysfunction and dementia, while endothelial dysfunction compromises cerebral blood flow, the blood-brain barrier and renal perfusion. Again, LVH from elevated combination waveform pressure leads to diastolic dysfunction and heart failure. Thus, elevated pulse wave velocity (PWV)and central aortic pulse augmentation indices are independent predictors of CAD, stroke, renal dysfunction, and all-cause mortality. (1) It is responsible for the rising risk of myocardial insufficiency, ischemia, LVH, and heart failure, cerebrovascular insufficiency or injury as well as renal injury and impairment with vascular aging.

The rate of vascular aging is multifactorial, including genetic susceptibilities as well as acceleration from vascular disease such as hypertension, atherosclerosis and diabetes. Recent trials have shown ACE inhibitors, angiotensin II blocks (ARBs) and Ca++ channel blockers have favorable effects on central aortic compliance, reducing LVH and reducing the risk of heart failure, stroke and renal impairment. In contrast, Beta blockers enhance central aortic BP augmentation by lengthening LV ejection time. Thus the reflected pulse waves arrive during late systole, augmenting the combined central aortic wave amplitude and LV workload.

Pulse wave velocity (PWV)has become a very good measure of aortic stiffness. PWV rises from 6m/sec in a young person to 10m/sec in a 65 y/o. It increases 2-fold from 20-80 y/o, due to a 4-fold reduction in aortic distensibility. (3) The CAFE study showed significant reduction in central artic BP and adverse cardiovascular events as well as renal impairment with Ca++ channel blockers, but not with atenolol plus thiazide Rx. (4) The REASON study showed ARBs reduced vascular stiffness, wave reflections, central aortic pulse pressure, vascular resistance, remodeling and thickness of resistance vessels. (5) Method/Design: The study will be human subject non-randomized observational study. This study will enroll approximately 500 patients. This was determined by a preliminary analysis of 140 patients, of which 19 had adverse cardiovascular events, within a week after surgery. The results of this preliminary study found average PWV was significantly higher in patients who developed postoperative cardiovascular events compared with patients who had uneventful postoperative course. (p-value 0.024). Therefore it was determined that 500 patients should be sufficient to see a statistically significant difference if there is one. This study will be conducted at day of surgery administration area and main operation room at University of Iowa Hospitals and clinics. Arterial stiffness will be measured at day of surgery administration area prior to the surgery. Carotid-Femoral Pulse Wave Velocity (Aortic Stiffness).

Carotid-femoral pulse wave velocity (cfPWV) will be determined by applanation tonometry using the Sphygmocor system by sequentially recording ECG-gated carotid and femoral artery waveforms. Pulse wave signals will be recorded by tonometers positioned at the base of the right common carotid artery and over the right femoral artery. The time (t) between the feet of simultaneously recorded waves will be determined as the mean of 10 consecutive cardiac cycles. PWV is calculated by the system software from the distance between measurement points (D) and the measured time delay (t) as follows: cfPWV = D/Δt (m/ s) where D is distance in meters and t is the time interval in seconds.

After consent, the subject will be taken to a private exam room where a noninvasive study of PWV and central aortic BP will be performed in supine position using the SphygmoCor sensor positioned over the carotid and femoral or radial artery pulse waveform, along with 3-lead EKG for QRS timing of the onset of systole. The SphygmoCor pulse wave sensor will be calibrated with an upper arm sphygmomanometer cuff BP. The vascular aging measurements will not be used to guide or alter medical decision making in the study. The study will take approximately 30 min. They will also not be repeated for this protocol either during or after surgery.

Pre and intraoperative data collection will include: ASA status, history of peripheral vascular disease, history of ischemic vascular disease, history of congestive heart failure, and history of cerebrovascular disease, intraop: all of the routine vital signs, anesthetic drug details, fluids, blood loss, and urine output data relevant to the surgical procedure. Any significant clinical AEs such as brady- or tachycardia (HR <50 or >100 for >10 min), hyper- or hypotension (BP >30% above or > 30% below awake), EKG rhythm or ST segment abnormality, abnormal BIS (anesthetic depth) or other EEG issue during anesthesia or surgery, and wake up difficulty will be documented in the clinical anesthesia electronic record. All other relevant monitoring data such as hypoxemia (pulse oximeter), hypo-or hyperventilation (capnography or arterial blood gas values) will be recorded in a clinical data file for each subject.

Postoperative data collection will include vital signs and any clinical cardiac, neurological or renal adverse events or other complications especially for the first 30 days, and any later events including all-cause mortality up to one year after surgery. Postoperative outcome information will be primarily collected via the medical record review. We do not plan to visit study subjects at bedside while recovering from surgery as inpatients, and will not schedule additional outpatient research follow up visits. However we also plan to call enrolled subjects at 1, 6, and 12 months after surgery to ask them whether they have experienced postoperative complications such as a a stroke, myocardial infarction, dysrhythmia such as atrial fibrillation, heart failure, respiratory failure, kidney function problem, renal failure or death.

ELIGIBILITY:
Inclusion Criteria:

Elective major surgery (scheduled > 4hours) patients, age 40 and up, will be recruited.

1. Surgical procedures and conditions that would meet INCLUSION criteria:

   1. GENERAL SURGERY- cholecystectomy, esophagectomy, gastric or bowel resection, gastric sleeve resections, liver resection, pancreatectomy, pheochromocytoma excision;
   2. HEAD & NECK SURGERY- laryngectomy radical neck dissection;
   3. NEUROSURGERY- craniotomy for brain tumor resection;
   4. ORTHOPEDIC SURGERY- total hip, total knee, total shoulder repair;
   5. SPINE SURGERY- multilevel lumbar or thoracic laminectomy, spinal stenosis decompression and stabilization;
   6. THORACIC SURGERY- open lobectomy, pneumonectomy
   7. UROLOGY- cystoprostatectomy, nephrectomy, and prostatectomy
   8. VASCULAR SURGERY- carotic endarterectomy, endovascular or open AAA repair, aortofemoral bypass, axillo-femoral bypass;
   9. GYNECOLOGY SURGERY- hysterectomy
2. At least ONE readily palpable CAROTID, RADIAL and FEMORAL artery pulse;
3. A signed informed consent form

Exclusion Criteria:

1. Cardiac surgery
2. Emergency surgical procedure;
3. Poorly or nonpalpable carotic, radial and/or femoral pulses;
4. A history of dizziness or fainting from carotic artery palpation
5. Atrial fibrillation or flutter

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing surgery and aged 40 and above
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2015-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Comparison of vascular stiffness between patients who develop a postoperative adverse cardiac event and those who don't | One month after surgery
  The study is aimed to compare arterial stiffness between patients who develop postoperative adverse cardiac complications and those who don't in patients who are undergoing major elective surgery. This includes coronary artery disease, congestive heart failure, cereberal artery disease, thrombolic event, carotid artery disease, kidney injury, valvular disease, significant EKG changes, respiratory failure and death. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)

SECONDARY OUTCOMES:
Comparison of vascular stiffness between patients who develop a postoperative adverse cardiac event and those who don't | 7 days
  The study is aimed to compare arterial stiffness between patients who develop postoperative adverse cardiac complications and those who don't in patients who are undergoing major elective surgery. This includes coronary artery disease, congestive heart failure, cerebral artery disease, thrombolic event, carotid artery disease, kidney injury, valvular disease, significant EKG changes, respiratory failure and death. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)
Comparison of vascular stiffness between patients who develop a postoperative adverse cardiac event and those who don't | 6 months
  The study is aimed to compare arterial stiffness between patients who develop postoperative adverse cardiac complications and those who don't in patients who are undergoing major elective surgery. This includes new onset from 6 month coronary artery disease, congestive heart failure, cerebral artery disease, thrombolic event, carotid artery disease, kidney injury, valvular disease, significant EKG changes, respiratory failure and death. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)
Comparison of vascular stiffness between patients who develop a postoperative adverse cardiac event and those who don't | 1 year
  The study is aimed to compare arterial stiffness between patients who develop postoperative adverse cardiac complications and those who don't in patients who are undergoing major elective surgery. This includes coronary artery disease, congestive heart failure, cerbral artery disease, thrombolic event, carotid artery disease, kidney injury, valvular disease, significant EKG changes, respiratory failure and death. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Background] Barodka VM, Joshi BL, Berkowitz DE, Hogue CW Jr, Nyhan D. Review article: implications of vascular aging. Anesth Analg. 2011 May;112(5):1048-60. doi: 10.1213/ANE.0b013e3182147e3c. Epub 2011 Apr 7. PMID 21474663
- [Background] HARKNESS ML, HARKNESS RD, MCDONALD DA. The collagen and elastin content of the arterial wall in the dog. Proc R Soc Lond B Biol Sci. 1957 Jun 25;146(925):541-51. doi: 10.1098/rspb.1957.0029. No abstract available. PMID 13441679
- [Background] O'Rourke MF, Nichols WW. Aortic diameter, aortic stiffness, and wave reflection increase with age and isolated systolic hypertension. Hypertension. 2005 Apr;45(4):652-8. doi: 10.1161/01.HYP.0000153793.84859.b8. Epub 2005 Feb 7. No abstract available. PMID 15699456
- [Background] Williams B, Lacy PS, Thom SM, Cruickshank K, Stanton A, Collier D, Hughes AD, Thurston H, O'Rourke M; CAFE Investigators; Anglo-Scandinavian Cardiac Outcomes Trial Investigators; CAFE Steering Committee and Writing Committee. Differential impact of blood pressure-lowering drugs on central aortic pressure and clinical outcomes: principal results of the Conduit Artery Function Evaluation (CAFE) study. Circulation. 2006 Mar 7;113(9):1213-25. doi: 10.1161/CIRCULATIONAHA.105.595496. Epub 2006 Feb 13. PMID 16476843
- [Background] London GM, Asmar RG, O'Rourke MF, Safar ME; REASON Project Investigators. Mechanism(s) of selective systolic blood pressure reduction after a low-dose combination of perindopril/indapamide in hypertensive subjects: comparison with atenolol. J Am Coll Cardiol. 2004 Jan 7;43(1):92-9. doi: 10.1016/j.jacc.2003.07.039. PMID 14715189
- [Background] Lee TH, Marcantonio ER, Mangione CM, Thomas EJ, Polanczyk CA, Cook EF, Sugarbaker DJ, Donaldson MC, Poss R, Ho KK, Ludwig LE, Pedan A, Goldman L. Derivation and prospective validation of a simple index for prediction of cardiac risk of major noncardiac surgery. Circulation. 1999 Sep 7;100(10):1043-9. doi: 10.1161/01.cir.100.10.1043. PMID 10477528
- [Background] Gupta PK, Gupta H, Sundaram A, Kaushik M, Fang X, Miller WJ, Esterbrooks DJ, Hunter CB, Pipinos II, Johanning JM, Lynch TG, Forse RA, Mohiuddin SM, Mooss AN. Development and validation of a risk calculator for prediction of cardiac risk after surgery. Circulation. 2011 Jul 26;124(4):381-7. doi: 10.1161/CIRCULATIONAHA.110.015701. Epub 2011 Jul 5. PMID 21730309
- See also: Related Info — http://www.surgicalriskcalculator.com/miorcardiacarrest